CLINICAL TRIAL: NCT00602108
Title: Phase II Study of Intra-operative Electron Irradiation and Hypofractionated External Beam Irradiation After Lumpectomy in Patients With Stage T1N0M0 or T2N0M0 Breast Cancer
Brief Title: Radiation Therapy in Treating Women Undergoing Lumpectomy for Stage I or Stage IIA Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William Wailing Wong, M.D., Mayo Clinic Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000583007; P30CA015083 (NIH); MCS314 (Other: Mayo Clinic Cancer Center); 806-04 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-01-23; First posted 2008-01-28 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: hypofractionated radiation therapy
Radiation: intraoperative radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving intraoperative radiation therapy after lumpectomy followed by external-beam radiation therapy may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects and how well radiation therapy works in treating women undergoing lumpectomy for stage I or stage IIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility and acute patient tolerance of intraoperative electron irradiation (IOERT) and hypofractionated external-beam irradiation (HYPORT) after lumpectomy for patients with stage I-IIA breast cancer treated with breast conservation therapy.
* To determine the local tumor control and distant tumor control rates for patients with stage I-IIA breast cancer treated with breast conservation therapy using IOERT and HYPORT after lumpectomy.
* To determine the long-term side effects and cosmetic outcome of IOERT to tumor bed and HYPORT after lumpectomy for patients with stage I-IIA breast cancer.

OUTLINE: Patients undergo lumpectomy per standard procedures. Patients undergo intraoperative electron irradiation (IOERT) to the tumor bed right after completion of lumpectomy with axillary lymph node dissection or sentinel lymph node biopsy.

Beginning 2-6 weeks after lumpectomy with axillary lymph node dissection/sentinel lymph node sampling and IOERT, patients receive hypofractionated external-beam irradiation once daily for 16 days.

After completion of study treatment, patients are followed at 3 months, every 6 months for 5 years, and then annually thereafter for 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary invasive breast carcinoma

  * Stage I-IIA disease (T1, N0, M0 or T2, N0, M0)
  * Pathologically determined single, discrete, and well-defined primary tumor ≤ 5 cm in diameter

    * Pathologically negative surgical margins
* No multicentric disease and/or diffuse malignant appearing microcalcifications

  * Micro-calcifications must be focal

    * Specimen radiograph is required after lumpectomy for tumors associated with malignant appearing calcifications to assure removal of all malignant appearing calcifications
    * Specimen radiograph is optional if the tumor appears as a discrete mass on mammogram
* No axillary lymph node involvement
* No evidence of metastatic breast cancer
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Menopausal status not specified
* No pre-existing collagen vascular disease except rheumatoid arthritis that does not require immunosuppressive therapy
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No prior irradiation to the area of planned radiation field
* No prior placement of breast prosthesis in the treated breast
* Concurrent hormonal therapy with external-beam irradiation allowed

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Toxicity: Up to 3 months post external beam radiation therapy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William W. Wong, MD, Study Chair — Mayo Clinic